CLINICAL TRIAL: NCT05708274
Title: The Role of Pharmacological Agents in Restoring Neuronal Excitability After Chronic Spinal Cord Injury (SCI)
Brief Title: Pharmacological Agents for Chronic Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lynda M. Murray, Assistant Professor, Bronx VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JJPVAMC IRB 1685818
Record Dates: First submitted 2022-12-27; First posted 2023-02-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
Keywords: Transcranial magnetic stimulation; Pharmacological agents; Transcutaneous spinal cord stimulation; Hand exercise
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Carboxypeptidase H

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, single-dose, randomized crossover investigation to one of four conditions: 1) CPH + hand training; 2) CD-LD + hand training; 3) ATX + hand training; and 4) placebo + hand training, performed at least a week apart. Outcomes measures will be assessed before and 60 minutes after study drug administration.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- CPH + hand training (Experimental): A single dose of Cyproheptadine (CPH) (8 mg) will be administered. Supplied as 2 over-encapsulated pills of 4 mg each.
  Interventions: Drug: CPH + hand training
- CD-LD + hand training (Experimental): A single dose of IR Carbidopa-levodopa (CD-LD) (50/200 mg) will be administered. Supplied as 2 over-encapsulated pills (25 mg carbidopa / 100 mg levodopa each).
  Interventions: Drug: CD-LD + hand training
- ATX + hand training (Experimental): A single dose of Atomoxetine (ATX) (40 mg) will be administered. Supplied as 1 over-encapsulated pill of 40 mg plus 1 placebo capsule.
  Interventions: Drug: ATX + hand training
- Placebo + hand training (Placebo Comparator): A single dose of Placebo will be administered. Supplied as 2 gelatin capsules, identical in number, size, shape and color, filled with microcrystalline cellulose.
  Interventions: Drug: Placebo + hand training

INTERVENTIONS:
Drug: CPH + hand training — Following a 10-minute rest after baseline measurements a single dose pharmacological agent or placebo will be administered, in blinded fashion, with up to 180 mL of noncarbonated water, on an empty stomach (minimum 2 hours without food). After capsule ingestion, participants will spend 50 minutes performing hand task-oriented training, resting for 10 minutes before undertaking post-intervention outcome measurements.
  Arms: CPH + hand training
Drug: CD-LD + hand training — Following a 10-minute rest after baseline measurements a single dose pharmacological agent or placebo will be administered, in blinded fashion, with up to 180 mL of noncarbonated water, on an empty stomach (minimum 2 hours without food). After capsule ingestion, participants will spend 50 minutes performing hand task-oriented training, resting for 10 minutes before undertaking post-intervention outcome measurements.
  Arms: CD-LD + hand training
Drug: ATX + hand training — Following a 10-minute rest after baseline measurements a single dose pharmacological agent or placebo will be administered, in blinded fashion, with up to 180 mL of noncarbonated water, on an empty stomach (minimum 2 hours without food). After capsule ingestion, participants will spend 50 minutes performing hand task-oriented training, resting for 10 minutes before undertaking post-intervention outcome measurements.
  Arms: ATX + hand training
Drug: Placebo + hand training — Following a 10-minute rest after baseline measurements a single dose pharmacological agent or placebo will be administered, in blinded fashion, with up to 180 mL of noncarbonated water, on an empty stomach (minimum 2 hours without food). After capsule ingestion, participants will spend 50 minutes performing hand task-oriented training, resting for 10 minutes before undertaking post-intervention outcome measurements.
  Arms: Placebo + hand training

SUMMARY:
The purpose of this study is to investigate the short-term effects of 3 approved FDA drugs (cyproheptadine (CPH), carbidopa-levodopa (CD-LD), and atomoxetine (ATX)) on motor responses when delivered in combination with hand training exercises in people with chronic spinal cord injury. The goal is to learn how to better strengthen connections between the brain and spinal cord after spinal cord injury, and if this connection is improved by one(or more) of the drugs. Multiple aspects of nerve transmission and muscle response will be measured via noninvasive brain and spinal cord stimulation, along with motor performance (dexterity and strength).

DETAILED DESCRIPTION:
Research will take place at the James J. Peters VA Medical Center (JJPVAMC), Bronx, NY. There are seven visits in total, including an initial evaluation and clinical assessment session. Each visit will last roughly 5 hours or less. We plan to enroll 28 participants with spinal cord injury over a two-year period.

The study is designed as a double-blind, placebo-controlled, single-dose, randomized crossover investigation involving four study drug visits (CPH, CD-LD, ATX, or placebo).

The same participants will partake in all four interventions in randomized order with at least 1-week washout representative of greater than 5x drug half-life; to avoid accumulative effects. To reduce potential learning effects from motor training and task-related outcome measurements, participants will partake in two motor training practice sessions prior to commencing the experiments for task familiarity.

This study will consist of electromyography (surface recordings of muscle activity), peripheral nerve stimulation, transcranial magnetic brain stimulation (TMS), and transcutaneous electrical spinal cord stimulation (TSCS), targeting the hand/arm muscles.

Though it is unlikely given the single-dose nature, participants may experience side effects following drug administration. Prior to consenting, all volunteers will undergo a comprehensive pre-screening evaluation including blood tests to ensure there are no contraindications.

Please note, there is no expectation of long-term benefit from this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age; clinically stable chronic (> 12 months) SCI at or above C8 spinal segment;
* Motor-incomplete with a score of 2 or more (out of 5) on manual muscle testing (MMT) of finger extension, finger flexion, or finger abduction in left or right hand(s); or able to perform thumb-index finger pinch of the left or right hand;
* Detectable stimulation-evoked muscle responses of the left or right first dorsal interosseous (FDI) and/or abductor pollicis brevis (APB); Detectable FDI/APB surface electromyography (EMG) muscle activity during thumb-index finger pinch;
* Must have stable: medication [≥ 30 days prior]; rehabilitation regimen [≥ 15 days prior];
* Must be able to: abstain from alcohol, smoking and caffeine consumption on the day prior/of each experiment; abstain from recreational drugs for the entirety of the study; commit to study requirements (i.e., 7 visits); provide informed consent.

Exclusion Criteria:

* History of moderate or severe head trauma (loss of consciousness for greater than one hour or evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging);
* History of other serious central or peripheral neurological injury;
* History of implanted brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants in the head (except inside mouth); cochlear implants; cardiac pacemaker/defibrillator; intracardiac lines; currently increased intracranial pressure; or other contraindications to brain stimulation or task performance;
* Ventilator dependence or patent tracheostomy site;
* Unstable syrinx, or multiple spinal cord lesions;
* Unclear diagnosis; History of stroke, brain tumor, brain abscess, or multiple sclerosis;
* Personal history of seizures; extensive family history of seizures; use of medications that lower seizure threshold (e.g., amphetamines, dalfampridine, and bupropion);
* Use of the study medications; Use of medications known to have significant adverse interactions with the study medication as described in the manufacturers' prescribing information [14 days prior]; previous allergic reaction or hypersensitivity to study drug(s);
* Presence of a medical condition that represents a risk for study drug(s) administration; evidence of liver disease or clinical jaundice; neutropenia; glaucoma; gastrointestinal ulcer(s); active malignancy; undiagnosed skin lesions; autoimmune disorders; chronic infectious diseases (e.g. HIV, hepatitis B or C); pregnancy or nursing mothers (a pregnancy urine test may be warranted); neurologic disorders (including a history of serious head trauma or seizures), and uncontrolled cardiovascular, metabolic, pulmonary or renal disease; premorbid, ongoing major depression or psychosis, altered cognitive status; bipolar disorder; suicidal ideation or past suicide attempts;
* History of severe hearing problems, loss or tinnitus;
* Presence of urinary infection, fever, pressure ulcer; or open skin lesions (shoulders or arms);
* Recent history (< 6 months) of recurrent autonomic dysreflexia, defined as a syndrome of sudden rise in systolic pressure greater than 20 mm Hg or diastolic pressure greater than 10 mm Hg, without rise in HR, accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, and blurry vision (closely monitored during all testing procedures);
* Heavy alcohol consumption (greater than equivalent of 5 oz of liquor) within previous 48 hours;
* Recent history (>1 year) of chemical substance dependency or significant psychosocial disturbance;
* Study participation of an investigational drug or device [60 days prior];
* Unsuitable for study participation as determined by the study physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Assessing task performance (dexterity) | Assess change from baseline to 10 minutes after completion of drug+task training.
  Unilateral manual dexterity will be assessed using the 9-Hole Peg Test (Aim 1a).

SECONDARY OUTCOMES:
Assessing task performance (dexterity) | Assess change from baseline to 10 minutes after completion of drug+task training.
  Unilateral manual dexterity will be assessed using the Box and Block Test (Aim 1a).
Assessing volitional grip strength | Assess change from baseline to 10 minutes after completion of drug+task training.
  Maximal grip force will be measured (Aim 1b). The attempt with the highest value will be used for analysis.
Assessing volitional pinch strength | Assess change from baseline to 10 minutes after completion of drug+task training.
  Maximal pinch force will be measured (Aim 1b). The attempt with the highest value will be used for analysis.
Assessing corticospinal plasticity | Assess change from baseline to 10 minutes after completion of drug+task training.
  Corticospinal plasticity will be measured via single-pulse TMS recruitment curves (Aim 2a).
Assessing cortical plasticity | Assess change from baseline to 10 minutes after completion of drug+task training.
  Short intracortical inhibition (SICI) and intracortical facilitation (ICF) will be evoked with paired-pulse TMS at various interstimulus intervals according to the methods previously employed (Murray & Knikou, 2017).
Assessing spinal plasticity | Assess change from baseline to 10 minutes after completion of drug+task training.
  Spinal plasticity will be measured via single-pulse TSCS recruitment curves (Aim 2b).
Tracking cardiovascular responses (heart rate) | Measured every 5-10 minutes, for up to 4 hours. Change will be compared to baseline.
  Observed measures of heart rate (HR) (Aim 3a) will be monitored throughout.
Tracking cardiovascular responses (blood oxygen saturation) | Measured every 5-10 minutes, for up to 4 hours. Change will be compared to baseline.
  Observed measures of blood oxygen saturation (SpO2) (Aim 3a) will be monitored throughout.
Tracking cardiovascular responses (blood pressure) | Measured every 5-10 minutes, for up to 4 hours. Change will be compared to baseline.
  Observed measures of blood pressure (BP) (Aim 3a) will be monitored throughout.
Tracking symptoms | Measured every 5-10 minutes, for up to 4 hours. Change will be compared to baseline.
  Participant-reported safety questionnaire (Aim 3b) will be monitored for any symptoms felt throughout the study.
Tracking side effects (drug administration) | Assess change from end of day 1 testing to 24 hours after study completion.
  Adverse event (AE) questionnaire (Aim 3b) related to any participant-reported experience following drug administration.
Tracking side effects (study testing stimulation) | Assess change from end of day 1 testing to 24 hours after study completion.
  Adverse event (AE) questionnaire (Aim 3b) related to any participant-reported experience following brain and/or spinal stimulation received during the experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda M Murray, PhD, Principal Investigator — Bronx VA Medical Center / James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters Veterans Affairs Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, individual-level data will be deposited to appropriate public repositories, such as Open Data Commons for Spinal Cord Injury (https://scicrunch.org/odc-sci), Figshare, or others.
  This will allow more powerful meta-analysis of disparate smaller studies, a need which is even more urgent in neurorehabilitation than in other fields that are more amenable to large drug studies.
Supporting Information: Study Protocol, SAP
Time Frame: Within 6 months of manuscript preparation.
Access Criteria: Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions described in the authorization and consent.
  A Data Use Agreement (DUA) will indicate adherence to any applicable Informed Consent provisions, and prohibits the recipient from identifying or re-identifying any individual whose data are included in the dataset.

DOCUMENTS (1):
  • Informed Consent Form (2025-11-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT05708274/ICF_000.pdf